CLINICAL TRIAL: NCT04083404
Title: Investigating Psychosocial Predictors & Employment Outcomes of Enhanced IPS Intervention A Prospective Cohort Study
Brief Title: Investigating Psychosocial Predictors & Employment Outcomes of Enhanced IPS Intervention
Status: Completed | Type: Observational
Sponsor: Queen Margaret University (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Susan Prior, Senior Research Fellow, Queen Margaret University
Other Study IDs: TS0001
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Psychiatric Disorder
Keywords: Complex mental health; employment; Enhanced Individual Placement & Support; Model of Human Occupation; Worker Role Interview
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this cohort study, using an existing database, is to seek to describe the relationship between psychosocial factors (independent variables) and employment outcomes (dependent variables) in a population of people with complex mental health problems receiving evidence-based supported employment (EBSE) augmented with theory-driven occupational therapy interventions. The intention is to understand the predictive nature of psychosocial factors on the positive outcome of success in achieving paid employment.

The Worker role interview (WRI) is routinely used in the research site; an National health Service (NHS) occupational therapy led vocational rehabilitation delivering EBSE service for people with complex mental health problems. An existing database of initial assessments and employment outcomes is available for investigation.

DETAILED DESCRIPTION:
The cohort study will be undertaken utilising a secondary dataset from an established vocational rehabilitation service (VRS). This service is experienced in providing intervention based on individual placement and support (IPS) with established high fidelity to the model. The team's interventions are also guided by the model of human occupation, (MOHO) and the Worker Role Interview is routinely completed with all patients accessing the service. The Worker Role Interview is a valid reliable measure of psychosocial items measuring of readiness for employment.

The consistency of intervention will be ensured as the service is routinely appraised for fidelity to the IPS by two experts, using a standardised assessment tool the IPS fidelity scale and the team has received ongoing training and regular caseload supervision to integrate evidence-based occupational therapy into practice. The experts appraising the service are independent of both the clinical service and the proposed research.

The established VRS provides an assessment and intervention for people with complex mental health problems. A dataset has been routinely collected over several years which is currently used to evaluate the service.

To address potential limitations of secondary data analysis the researcher has an established relationship with clinicians in the VRS and was involved in the selection of routine measures now used to evaluate the service. It is, therefore, possible to be confident that a consistent and standard dataset is available for analysis. Ongoing training and consultation have been provided by the researcher to the clinical service to ensure the data quality.

Data Collection The data will be managed and transferred by a trained researcher on site at both services.Data will be robustly anonymised prior to transfer. Data will be transferred from NHS secure network to secure network within Queen Margaret University using a secure email service approved by the Department of Health.

The dataset comprises; Research identification (ID) code Gender Age on Admission Ethnicity Marital Status Living situation (alone/shared/supported accommodation) Quintile range of Scottish Index of Multiple Deprivation Educational attainment Previous employment ICD10 Worker role interview items Date of assessment WRI Assesses Abilities & Limitations WRI Expectation of Success in Work WRI Takes Responsibility WRI Commitment to Work WRI Work-Related Goals WRI Enjoys Work WRI Pursues Interests WRI Appraises Work Expectations WRI Influence of Other Roles WRI Work Habits WRI Daily Routines WRI Adapts Routine to Minimize Difficulties WRI Perception of Physical Work Setting WRI Perception of Family and Peers WRI Perception of Boss and/or Company WRI Perception of Co-workers Employment goal Date of final goal review Outcome of goal (successful/ unsuccessful in attaining employment)

Sample; Based on the guideline of a minimum of 10 events per predictor variable, a sample size of 200 would allow for the robust estimation of 8 variables in the model.

Analysis Plan The collected data will be subject to analysis with the use of multiple logistic regression using the R data analysis software. Multiple logistic regression will allow the construction of models which examine the effects of psychosocial predictors on the probability of a person with complex mental health problems attaining paid employment. Possible confounds which may influence outcomes will be controlled for (e.g. age, gender, educational achievement, history of employment). Interpretation of the analysis will be shared and discussed with clinicians who are expert in their field to ensure that findings are considered from both a statistical significance and clinical significance position.

ELIGIBILITY:
Inclusion Criteria:

* self-referred to vocational rehabilitation service
* goal of open paid employment or education
* supported by community mental health teams
* capacity to consent

Exclusion Criteria:

* Lack capacity for informed consent.
* Refusal or withdrawal of informed consent
* Incomplete initial assessment data
* Withdrawal from participation in service prior to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complex mental health problems; unemployed
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Forsyth, PhD, Study Director — Queen Margaret University

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

REFERENCES:
- [Background] Kinoshita Y, Furukawa TA, Kinoshita K, Honyashiki M, Omori IM, Marshall M, Bond GR, Huxley P, Amano N, Kingdon D. Supported employment for adults with severe mental illness. Cochrane Database Syst Rev. 2013 Sep 13;2013(9):CD008297. doi: 10.1002/14651858.CD008297.pub2. PMID 24030739
- [Background] Bond GR, Peterson AE, Becker DR, Drake RE. Validation of the Revised Individual Placement and Support Fidelity Scale (IPS-25). Psychiatr Serv. 2012 Aug;63(8):758-63. doi: 10.1176/appi.ps.201100476. PMID 22660842
- [Background] Forsyth K, Braveman B, Kielhofner G, Ekbladh E, Haglund L, Fenger K, Keller J. Psychometric properties of the Worker Role Interview. Work. 2006;27(3):313-8. PMID 17006008
- [Derived] Prior S, Maciver D, Aas RW, Kirsh B, Lexen A, van Niekerk L, Irvine Fitzpatrick L, Forsyth K. An enhanced individual placement and support (IPS) intervention based on the Model of Human Occupation (MOHO); a prospective cohort study. BMC Psychiatry. 2020 Jul 8;20(1):361. doi: 10.1186/s12888-020-02745-3. PMID 32641009

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Individual Placement and Support (IPS) Programme: An enhanced individual placement and support (IPS) intervention based on the Model of Human Occupation
Period: Overall Study
Arm/Group | Enhanced Individual Placement and Support (IPS) Programme
Started | 202
Completed | 202
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enhanced IPS Programme: An enhanced individual placement and support (IPS) intervention based on the Model of Human Occupation
Arm/Group | Enhanced IPS Programme
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 185
  Ethnicity: Other ethnic group | 17
Marital Status [Count of Participants; unit: Participants]
  Married / de facto relationship | 33
  Single | 163
  missing data | 6
Social Situation [Count of Participants; unit: Participants]
  living with others | 97
  living alone | 101
  missing data | 4
Scottish Indices of Multiple Deprivation [Count of Participants; unit: Participants] — The Scottish Index of Multiple Deprivation is the Scottish Government's official tool for identifying areas in Scotland concentrations of deprivation by incorporating several different aspects of deprivation (multiple-deprivations) and combining them into a single index.
  Counts of participants living in each quintile are provided, from the most deprived 20% to the least deprived 20%.
  Participants
    most deprived quintile 1 | 38
    quintile 2 | 35
    quintile 3 | 33
    quintile 4 | 32
    least deprived quintile 5 | 64
Educational Attainment [Count of Participants; unit: Participants]
  Did Not Attain School Quals | 18
  Exams from School | 61
  Further Education | 121
  missing data | 2
Previous Employment [Count of Participants; unit: Participants]
  Previous employment | 182
  No previous employment | 20
ICD10 [Count of Participants; unit: Participants] — The International Classification of Diseases defines the universe of diseases, disorders, injuries and other related health conditions. Complex mental health conditions experienced by participants of this study were classified under the categories ICD F2; Schizophrenia, schizotypal, delusional, and other non-mood psychotic disorders. And ICD F3; Mood [affective] disorders. Or ICD other.
  Participants
    ICD10 F2 | 105
    ICD10 F3 | 67
    ICD10 other | 30
Worker Role Interview Item Assesses Abilities and Limitations [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Assesses Abilities and Limitations is defined as the individual's capacity to accurately assess his/her abilities and what they mean for work performance (Braveman et al 2005).
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 35
    Supports | 102
    Interferes | 59
    Strongly interferes | 5
    Missing data | 1
Worker Role Interview Item Expectation of job success [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Expectation of Success in Work: a client's belief that he/she will be able to work. Overall, raters are guided to consider the general degree of optimism the person has about working.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 17
    Supports | 92
    Interferes | 88
    Strongly interferes | 5
    Missing data | 0
Worker Role Interview Item Takes Responsibility [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Takes Responsibility: how much responsibility a client takes for his/her work actions and their consequences.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 30
    Supports | 81
    Interferes | 82
    Strongly interferes | 9
    Missing data | 0
Worker Role Interview Item Commitment to work [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Commitment to Work: Defined as a client's commitment to work and importance placed on work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 69
    Supports | 106
    Interferes | 27
    Strongly interferes | 0
    Missing data | 0
Worker Role Interview Item Work-related goals [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Work-Related Goals: Defined as the client's ability to set and attain goals at his/her work setting.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 29
    Supports | 89
    Interferes | 74
    Strongly interferes | 9
    Missing data | 1
Worker Role Interview Item Enjoys work [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Enjoys Work: Defined as the pleasure or enjoyment client finds within work. Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 36
    Supports | 114
    Interferes | 42
    Strongly interferes | 5
    Missing data | 5
Worker Role Interview Item Pursues interests [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Pursues Interests: the ability of an individual to assess his/her own interests and find ways to use these skills in and/or outside of the work situation.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 32
    Supports | 77
    Interferes | 81
    Strongly interferes | 10
    Missing data | 2
Worker Role Interview Item Appraises work expectations [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Appraises Work Expectations: ability to internalize both general and specific expectations of work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 50
    Supports | 108
    Interferes | 34
    Strongly interferes | 6
    Missing data | 4
Worker Role Interview Item Influence of other roles [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Influence of Other Roles: Defined as how much other roles in the client's life influence his/her return to work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 50
    Supports | 96
    Interferes | 54
    Strongly interferes | 2
    Missing data | 0
Worker Role Interview Item Work Habits [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Work Habits: Defined as the degree of organization and routine in work. Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 33
    Supports | 96
    Interferes | 52
    Strongly interferes | 16
    Missing data | 5
Worker Role Interview Item Daily Routine [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Daily Routine: Defined as the degree of organization and routine outside of work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 13
    Supports | 62
    Interferes | 106
    Strongly interferes | 20
    Missing data | 1
Worker Role Interview Item Adapts routines to minimize difficulties [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Adapts Routines to Minimize Difficulties: Defined as how the person has managed use of time, routine, and habits since the injury or since being out of work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 13
    Supports | 87
    Interferes | 85
    Strongly interferes | 16
    Missing data | 1
Worker Role Interview Item Perception of physical work setting [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Perception of Physical Work Setting: The client's impression of how a work environment may support or hinder his/ her return to work or finding and keeping work Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 27
    Supports | 107
    Interferes | 46
    Strongly interferes | 2
    Missing data | 20
Worker Role Interview Item Perception of family and peers [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Perception of Family and Peers: Defined as the influence family's and peers' have on the client's ability to return to previous work Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 50
    Supports | 92
    Interferes | 33
    Strongly interferes | 11
    Missing data | 16
Worker Role Interview Item Perception of boss and/or company [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Perception of Boss and/or Company: Defined as the influence of boss and/or company on the ability of client to return to previous work or find and keep work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 26
    Supports | 52
    Interferes | 57
    Strongly interferes | 9
    Missing data | 58
Worker Role Interview Item Perception of co-workers [Count of Participants; unit: Participants] — The worker role interview (WRI) (Braveman et al. 2005) is a semi-structured interview & rating scale identifying psychosocial factors that influence a client's ability to work. The WRI is a valid, reliable assessment tool, which can discriminate between levels of work status.
  Perception of Co-workers: Defined as co-workers' influence on client's ability to return to previous work and find and keep work.
  Clinicians determine if the item strongly supports; supports; interferes or strongly interferes with an individual's ability to work.
  Participants
    Strongly supports | 26
    Supports | 63
    Interferes | 40
    Strongly interferes | 8
    Missing data | 65

OUTCOME MEASURES:

1. Primary Outcome: Attainment of Employment or Education
Description: successful attainment of open employment or educational opportunity / unsuccessful
Time Frame: 1day
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced IPS Programme
Number analyzed (Participants) | 202
Participants
  Attained employment or education | 128
  Did not attain employment or education | 74

2. Other Pre Specified Outcome: Time to Attainment of Employment or Education
Description: Time to outcome for those successfully attaining employment or education
Time Frame: 1day-69months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Enhanced IPS Programme
Number analyzed (Participants) | 128
months | 8.435 [5.055 to 16.742]

ADVERSE EVENTS:
Time Frame: 1day to 69mths
Arm/Group | Enhanced IPS Programme
All-Cause Mortality (participants affected / at risk) | 0/202
Serious Adverse Events (participants affected / at risk) | 0/202
Other Adverse Events (participants affected / at risk) | 0/202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04083404/Prot_SAP_000.pdf